CLINICAL TRIAL: NCT03293992
Title: A Phase I, Multi-Center, Randomized, Adaptive, Investigator/Patient Masked, Multiple-Ascending Dose, Placebo and Active Comparator-Controlled Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7058584 Following 7 Days of Topical Instillation of Eye Drops in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7058584 Following 7 Days of Instillation of Eye Drops in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP39863
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Glaucoma, Open-angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.01% RO7058584 or Matching Placebo (Experimental)
  Interventions: Drug: 0.01% RO7058584; Drug: Matching Placebo
- 0.1% RO7058584 or Matching Placebo (Experimental)
  Interventions: Drug: 0.1% RO7058584; Drug: Matching Placebo
- 1% RO7058584 or Matching Placebo (Experimental)
  Interventions: Drug: 1% RO7058584; Drug: Matching Placebo
- RO7058584 and Latanoprost 0.005% (Experimental)
  Interventions: Drug: 0.01% RO7058584; Drug: 0.1% RO7058584; Drug: 1% RO7058584; Drug: Latanoprost 0.005%

INTERVENTIONS:
Drug: 0.01% RO7058584 — Once daily morning administration for 7 days
  Arms: 0.01% RO7058584 or Matching Placebo; RO7058584 and Latanoprost 0.005%
Drug: 0.1% RO7058584 — Once daily morning administration for 7 days
  Arms: 0.1% RO7058584 or Matching Placebo; RO7058584 and Latanoprost 0.005%
Drug: 1% RO7058584 — Once daily morning administration for 7 days
  Arms: 1% RO7058584 or Matching Placebo; RO7058584 and Latanoprost 0.005%
Drug: Matching Placebo — Once daily morning administration for 7 days
  Arms: 0.01% RO7058584 or Matching Placebo; 0.1% RO7058584 or Matching Placebo; 1% RO7058584 or Matching Placebo
Drug: Latanoprost 0.005% — Once daily morning or evening dosing
  Arms: RO7058584 and Latanoprost 0.005%

SUMMARY:
This is a Phase I, multi-center, randomized, adaptive, investigator/patient-masked, placebo-controlled, parallel multiple-ascending dose study (Part A) with an extension including up to two selected doses from Part A and latanoprost 0.005% as active comparator (Part B).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years of age inclusive, at the time of signing the informed consent form
* Confirmed diagnosis of ocular hypertension (OHT) or primary open-angle glaucoma (POAG) in both eyes as determined by the investigator at screening
* Treatment-naïve participants or participants who are able to safely stop their Intraocular pressure (IOP)-lowering medication(s) prior to randomization according to the required minimum washout periods
* At baseline visit, IOP ≥ 24 millimeters of mercury (mmHg) in the morning (8:00 AM ± 1h) and ≥ 22 mmHg in the afternoon (2:00 PM ± 1h) measurement in the same eye and ≤ 34 mmHg at all timepoints in both eyes
* Best corrected logarithm of the minimum angle of resolution (logMAR) visual acuity score of 0.7 or better in each eye as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity test at screening
* Central corneal thickness (pachymetry) measurement 450 to 620 micrometers (μm) in both eyes at screening
* Cup-to-disc ratio ≤ 0.8 (both eyes) at screening
* Anterior chamber angle is open and non-occludable (both eyes) as confirmed by the investigator by gonioscopy examination at screening

Exclusion Criteria:

* Advanced visual field defects
* Other forms of glaucoma than POAG or OHT
* Any abnormality preventing reliable applanation tonometry
* Any clinically significant corneal scarring, haze or opacity
* Uncooperativeness of the participant that restricts adequate examination of IOP, ocular fundus or anterior chamber
* Any presence or history of uveitis or other history of any ocular inflammatory disease.
* History or signs of penetrating ocular trauma
* Risk of visual field or visual acuity worsening in either eye as a consequence of glaucoma progression or consequence of participation in the trial or any other ocular disease, according to the investigator's best judgment
* History of any glaucoma surgery
* History of refractive surgery
* Any other intra-ocular surgery within six months of screening
* Any active ocular disease requiring treatment.
* Use of any listed prohibited medications
* Current enrollment or past participation within the last 30 days before the screening visit in any other clinical study involving an investigational study treatment or any other type of medical research
* Any participant who is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff thereof, directly involved in the conduct of the protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence, Severity, and Causal Relationship of Ocular and Systemic Adverse Events (AEs) | Up to 12 weeks
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Incidence of Abnormal Laboratory Findings | Up to 12 weeks
Incidence of Blood Pressure Abnormalities | Up to 12 weeks
Incidence of Pulse Rate Abnormalities | Up to 12 weeks
Incidence of Electrocardiogram (ECG) Findings | Up to 12 weeks
Change From Baseline in Mean Intraocular pressure (IOP) After 7 Days of Study Drug Administration | 7 days
  IOP will be assessed by Goldman Applanation tonometry.

SECONDARY OUTCOMES:
Change From Baseline in Mean Intraocular pressure (IOP) at Matched Clock-Times After 7 Days of Study Drug Administration | 7 days
  IOP will be assessed by Goldmann Applanation tonometry
Cmax of RO7058584 | Up to Day 8
  Cmax is the maximum observed plasma concentration.
Tmax of RO7058584 | Up to Day 8
  Tmax is the time to maximum observed plasma concentration.
Ctrough of RO7058584 | Up to Day 8
  Ctrough is the concentration at the end of a dosing interval before the next dose administration.
AUC0-24h of RO7058584 | Up to Day 8
  AUC0-24h is the area under the plasma concentration versus time curve (AUC) from Time 0 to 24 h post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - Arizona Eye Center, Chandler, Arizona
  - Sall Research Medical Center, Artesia, California
  - United Med Res Inst, Inglewood, California
  - Eye research foundation, Newport Beach, California
  - Rocky Mountain Lions Eye Inst, Aurora, Colorado
  - Eye Care Centers Management, Inc. (Clayton Eye Center), Morrow, Georgia
  - Coastal Research Associates, Roswell, Georgia
  - Texan Eye/Keystone Research, Austin, Texas